CLINICAL TRIAL: NCT02082834
Title: Post EVAR Endoleak Detection : Model-based Iterative Reconstruction (MBIR) vs Adaptive Statistical Iterative Reconstruction (ASIR) CTA; a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0184
Record Dates: First submitted 2014-02-21; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Post EVAR Endoleak Detection
Keywords: Endovascular aneurysm repair EVAR; Endoleak/diagnosis; VEOTM; Model-based iterative reconstruction (MBIR); Adaptive statistical iterative reconstruction (ASIR); Aortic Aneurysm; Low dose; Prospective; CTA
MeSH Terms: conditions — Endoleak; Disease; Aortic Aneurysm

ARMS (1):
- EVAR (Experimental)
  Interventions: Other: abdominal MDCT examination

INTERVENTIONS:
Other: abdominal MDCT examination

SUMMARY:
The purpose of the study is to compare the accuracy of the diagnosis of endoleak in patient with EVAR comparing Adaptive statistical iterative reconstruction (ASIR) CTA and Model-based iterative reconstruction (MBIR- VEO TM).

DETAILED DESCRIPTION:
Background:

The aortic aneurysm is a common and serious disease share its complications (rupture ) , often fatal. It is recognized that pass a certain diameter surgical or endovascular treatment reduces mortality by avoiding treatment in extreme provider of high morbidity and mortality emergency. Endovascular anevrysm repair (EVAR) treatment has proven effective but unfortunately this treatment presents complications ( endoleak ) should be sought systematically by repeated checks CT . The irradiation in these patients is a major problem with repeated exposure radiation. The follow up of these patients requires repeated CT because endoleaks can be delayed.

Iterative reconstruction of previous generation have reduced the dose , we dispose the last Model-based iterative reconstruction (" VEO " ) for a further reduction of patient dose . This technique has not yet been evaluated in the detection of endoleaks.

The purpose of the study is to compare conventional CTA (ASIR50) ( gold standard now) with Model-based iterative reconstruction (MBIR- VEO TM) in the detection ( and classification ) of endoleaks in patients traited by EVAR.

All patient admited in Radiology to follow up his EVAR is included in the study and receive both CT: Adaptive statistical iterative reconstruction (ASIR) CTA and Model-based iterative reconstruction (MBIR- VEO TM) and the result of thoses 2 CT are compared by 2 readers (blinded of the result) The BMI , other complications, the DLP , dose reduction and quality of the examination is noted .

ELIGIBILITY:
Inclusion Criteria:

* informed and a written consent
* all patients consulting to follow up his EVAR
* 18-90 years
* French

Exclusion Criteria:

* pregnant
* juvenile patients
* patient who refusal the study
* CI of contrast iodine injection : CI of ultravist
* llergy
* renal failure creatinemy <30 ml/min

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Presence or absence of endoleak after EVAR using CT evaluation | at day 1

SECONDARY OUTCOMES:
Type of endoleak, BMI (body mass index | at day 1
Diameter of the aneurysm | at day 1
Objective and subjective image quality | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean Cassagnes, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France